CLINICAL TRIAL: NCT01816360
Title: The Effects of Olfactory Aromatherapy and Yogatherapy Breathing Exercises on the Quality of Life, Stress Levels, Coping Strategies and Hot Flashes Intensity and Frequence in Climacteric Women
Brief Title: Aromatherapy and Yogatherapy for Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cassandra Santantonio de Lyra, MSc, Master in Science, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AromaYoga
Record Dates: First submitted 2013-03-18; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Menopause; Hot Flashes; Hot Flushes
Keywords: Womens health; Menopause; Complementary therapies; Aromatherapy; Essential oils; Yogatherapy; Psychoneuroendocrineimmunology
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aromatherapy group (Experimental): 20 sessions of olfactory aromatherapy using protocol.
  Interventions: Other: Olfactory aromatherapy
- Yogatherapy group (Experimental): 20 sessions of yogatherapy with aroma-placebo using protocol.
  Interventions: Other: Yogatherapy
- Aromatherapy-Yogatherapy group (Experimental): 20 sessions of yogatherapy with olfactory aromatherapy, using protocol.
  Interventions: Other: Olfactory aromatherapy; Other: Yogatherapy
- Control group (No Intervention): Control group in the waiting-list model (all volunteers were offered the treatment after the completion of data collection).

INTERVENTIONS:
Other: Olfactory aromatherapy — Inhalation of essential oils.
  Arms: Aromatherapy group; Aromatherapy-Yogatherapy group
Other: Yogatherapy — Yogatherapy respiratory exercises.
  Arms: Aromatherapy-Yogatherapy group; Yogatherapy group

SUMMARY:
The purpose of this study is to verify and analyse psychological and physiological effects of olfactory aromatherapy and yogatherapy respiratory exercises, together and separately, on the quality of life, levels of stress, quality of sleep and intensity and frequence of hot flashes in climacteric women.

DETAILED DESCRIPTION:
Introduction: Menopause is the period in which reproductive life ends and senescence begins. Because of the increase in life expectancy there are more women reaching this period. Although it is a physiological change, it is frequently accompanied by disagreeable symptoms that can influence quality of life and sleep in a negative manner. The most common symptom is hot flashes. The traditional treatment for the symptoms is hormone replacement therapy, that has many important side effects, such as increase in cancer incidence. This therapy also has dubious effects on psychosexual symptoms and quality of life. This justifies the study of other more secure treatments. Aromatherapy can be a particularly efficacious treatment for hot flashes because it has therapeutic mechanisms that are similar to the physiological mechanisms of hot flashes. It is also a secure therapy with little side effects, specially when applied in inhalation (olfactory aromatherapy). Yogatherapy can also influence psychoneuroedocrineimmunological axis similar to the physiological axis of hot flashes. Yogatherapy includes respiratory exercises that can potentiate the effects of olfactory aromatherapy. Because of this, it can be beneficial to apply aromatherapy and yogatherapy together. These therapies were studied as they are applied in clinical practice. The psychoneuroendocrineimmunological model permits the study of the effects of both these therapies aiming at increase in quality of life, from a psychosomatic and global point of view. The global approach is important in the study of menopause because it has both psychological and physiological characteristics. Objective: verify and analyse psychological and physiological effects of olfactory aromatherapy and yogatherapy respiratory exercises, together and separately, on the quality of life, levels of stress, quality of sleep and intensity and frequence of hot flashes in climacteric women. Material and methods: The study is a placebo-controlled double-blind clinical trial, with restrict randomization methods (that allow groups of the same size). Recruitment of voluntaries was made using posters and electronic messages in websites. Data was collected at the "Centro de Práticas Esportivas da Universidade de São Paulo" (Sport Centre of the University of Sao Paulo). The study will have four groups: aromatherapy, yogatherapy, both therapies and control-placebo group. Appraisal was done using questionnaires for personal data, social-economical data, stress levels, quality f sleep levels, body resonance levels, quality of life levels, climacteric influence on quality of life and physiological data (heart rate, breathing rate, blood pressure and body temperature). Appraisal was done before, during and after 20 treatment sessions. The research was approved by the "Comitê de Ética em Pesquisa da Escola de Educação Fisica e Esporte da Universidade de São Paulo" (Ethics Committee of the Sport and Physical Education School of the University of Sao Paulo). Data will be analysed using descriptive statistics, Student t-test, ANOVA variance analysis and Pearson correlation, considering significance levels of p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Age from 45 to 60 years
* Women who reported having hot flashes for at least 6 months

Exclusion Criteria:

* History of hysterectomy, oophorectomy or endometrial ablation
* Chemotherapy in the last 5 years
* Women receiving treatment for menopausal symptoms (including hormone replacement therapy)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in frequence and intensity of hot flashes | Before, after 10 sessions (5 weeks) and after 20 sessions (10 weeks) of intervention.
  Change in frequence and intensity of hot flashes using questionnaire developed for this study.

SECONDARY OUTCOMES:
Change in quality of sleep | Before, after 10 sessions (5 weeks) and after 20 sessions (10 weeks) of intervention.
  Change in quality of sleep using the Pittsburgh Index of Quality of Sleep, translated to portuguese.
Body resonance | Before intervention
  Body resonance using the "RESCORP" (ressonância corporal) brazilian questionnaire.
Psycho-social influences on the effects of the aroma. | Before, after 10 sessions (5 weeks) and after 20 sessions (10 weeks) of intervention.
  Influence of aroma preferences and olfactory memories in effects of aroma. Changes in aroma preferences. Using questionnaire developed for this study.
Personal data | Before intervention
  Personal data for evaluating possible correlations and verifying possible risk factors for climacteric symptoms.
Change in stress level | At beginning of study and after each session of intervention (twice a week for 10 weeks).
  Change in stress level throughout the whole 20 sessions of intervention, using the Visual Analogue Scale for Stress.
Change in quality of life | Before, after 10 sessions (5 weeks) and after 20 sessions (10 weeks) of intervention.
  Change in quality of life measured by the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra S Lyra, MSc, Principal Investigator — Doctoral student at Universidade de Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil